CLINICAL TRIAL: NCT05862610
Title: A Prospective, Randomized, Controlled Phase II Clinical Study of Trilaciclib Combined With Standard Treatment Project As a Neoadjuvant Treatment For Triple Negative Breast Cancer
Brief Title: The Study of Trilaciclib Combined With Chemotherapy On The Neoadjuvant Therapy of TNBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMA-BC-001
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Breast Neoplasm
Keywords: Trilaciclib/TNBC/Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — trilaciclib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trilaciclib plus chemotherapy (Trilaciclib+AC-T) (Experimental): Trilaciclib: 240mg/m2 IV d1,within 4h before chemotherapy epirubicin: 100mg/m2 IV d1,Q2W/Q3W (decided by researchers),4 cycles cyclophosphamide:600mg/m2 IV d1,Q2W/Q3W (decided by researchers),4 cycles albumin-bound paclitaxel:100mg/m2 IV d1,8,15,Q3W,4cycles
  Interventions: Drug: Trilaciclib plus chemotherapy
- Chemotherapy (AC-T) (Experimental): epirubicin: 100mg/m2 IV d1,Q2W/Q3W (decided by researchers),4 cycles cyclophosphamide:600mg/m2 IV d1,Q2W/Q3W (decided by researchers),4 cycles albumin-bound paclitaxel:100mg/m2 IV d1,8,15,Q3W,4cycles
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Trilaciclib plus chemotherapy — Trilaciclib: 240mg/m2 IV d1,within 4h before chemotherapy epirubicin: 100mg/m2 IV d1,Q2W/Q3W (decided by researchers),4 cycles cyclophosphamide:600mg/m2 IV d1,Q2W/Q3W (decided by researchers),4 cycles albumin-bound paclitaxel:100mg/m2 IV d1,8,15,Q3W,4cycles
  Other Names: Trilaciclib+AC-T
  Arms: Trilaciclib plus chemotherapy (Trilaciclib+AC-T)
Drug: Chemotherapy — epirubicin: 100mg/m2 IV d1,Q2W/Q3W (decided by researchers),4 cycles cyclophosphamide:600mg/m2 IV d1,Q2W/Q3W (decided by researchers),4 cycles albumin-bound paclitaxel:100mg/m2 IV d1,8,15,Q3W,4cycles
  Other Names: AC-T
  Arms: Chemotherapy (AC-T)

SUMMARY:
To evaluate the efficacy and safety of trilaciclib combined with standard treatment project as a neoadjuvant treatment for triple negative breast cancer

DETAILED DESCRIPTION:
Trilaciclib indication: Trilaciclib, a CDK4/6 inhibitor, was used before chemotherapy to reduce the incidence of bone marrow suppression and approved by the FDA for small cell lung cancer patients in 2021.

ELIGIBILITY:
Inclusion Criteria:

* Newly treated patients aged ≥ 18 years;
* ECOG score 0-1;
* Breast cancer meets the following standards:

  1. Histologically confirmed invasive breast cancer
  2. Tumor staging: cT2-4, cNany, cM0 or cT1, cN1-3, cM0;
* Hormone (estrogen and progesterone) receptor negative tumors confirmed by histological or cytological records (defined as nuclear staining rate<1% based on immunohistochemistry [IHC] evaluation) and Her-2 negative, non overexpressing tumors (based on IHC [0 or 1+] or in situ hybridization [ratio<2.0] or average Her-2 gene copy number<4 signals/nucleus);
* Within the first two weeks of the screening period, no G-CSF, TPO, IL-11, ESA, iron, platelet transfusion, or blood transfusion have been used.
* The functional level of the main organs must meet the following requirements:

  1. Blood routine: Neutrophils (ANC)≥1.5×109/L, platelet count (PLT)≥90×109/L, hemoglobin (Hb)≥90g/L
  2. Blood biochemistry: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN, serum creatinine (Cr)≤1.5×ULN, bilirubin<1.5 ULN;
* For female patients who have not undergone menopause or surgical sterilization: During the treatment period and at least 7 months after the last dose in the study treatment, consent to abstinence or use effective contraceptive methods.
* Volunteer join this study, sign an informed consent form, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

* Previously received anti-tumor treatment for any malignant tumor;
* Subjects who are unable to accept or tolerate preoperative chemotherapy due to various reasons;
* The patient has undergone major surgical procedures unrelated to breast cancer within 4 weeks before enrollment, or has not fully recovered from such surgical procedures;
* Serious heart disease or discomfort, including but not limited to the following diseases:

  1. A confirmed history of heart failure or systolic dysfunction (LVEF<50%);
  2. High risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate>100bpm, significant ventricular arrhythmias (such as ventricular tachycardia) or higher-level atrioventricular block (such as Mobitz II second degree atrioventricular block or third degree atrioventricular block);
  3. Angina pectoris requiring treatment with anti angina drugs;
  4. Heart valve disease with clinical significance;
  5. ECG shows transmural myocardial infarction;
  6. Poor control of hypertension (systolic blood pressure>180mmHg and/or diastolic blood pressure>100mmHg)
* Those with a known history of allergies to the drug components of this protocol;
* Breastfeeding female patients, those with fertility and positive baseline pregnancy test results, or those of childbearing age who are unwilling to take effective contraceptive measures during the entire trial period and within 7 months after the last study medication;
* Any other circumstances in which the researcher believes that the patient is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of CIN | From date of randomization until the date of surgery, assessed up to 6 months
  The incidence of ≥3 grade neutropenia

SECONDARY OUTCOMES:
The incidence of CIT | From date of randomization until the date of surgery, assessed up to 6 months
  The incidence of ≥3 grade thrombopenia
The incidence of CIA | From date of randomization until the date of surgery, assessed up to 6 months
  The incidence of ≥3 grade anemia
pCR rate | From date of randomization until the date of surgery, assessed up to 6 months.
  Rate of pCR using the definition of ypT0/Tis ypN0 as assessed by the local pathologist.
ORR | From date of randomization until the date of PD (up to 24 months)
  Objective Response Rate
OS | From date of randomization until the date of death(up to 24 months)
  Overall survival
DFS | From date of randomization until the date of toxicity or PD (up to 24 months)
  Disease-free survival
Adverse event | Frame:From date of randomization until the date of toxicity or PD (up to 24 months)
  Number of participants with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, Doc, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiss JM, Csoszi T, Maglakelidze M, Hoyer RJ, Beck JT, Domine Gomez M, Lowczak A, Aljumaily R, Rocha Lima CM, Boccia RV, Hanna W, Nikolinakos P, Chiu VK, Owonikoko TK, Schuster SR, Hussein MA, Richards DA, Sawrycki P, Bulat I, Hamm JT, Hart LL, Adler S, Antal JM, Lai AY, Sorrentino JA, Yang Z, Malik RK, Morris SR, Roberts PJ, Dragnev KH; G1T28-02 Study Group. Myelopreservation with the CDK4/6 inhibitor trilaciclib in patients with small-cell lung cancer receiving first-line chemotherapy: a phase Ib/randomized phase II trial. Ann Oncol. 2019 Oct 1;30(10):1613-1621. doi: 10.1093/annonc/mdz278. PMID 31504118
- [Background] Daniel D, Kuchava V, Bondarenko I, Ivashchuk O, Reddy S, Jaal J, Kudaba I, Hart L, Matitashvili A, Pritchett Y, Morris SR, Sorrentino JA, Antal JM, Goldschmidt J. Trilaciclib prior to chemotherapy and atezolizumab in patients with newly diagnosed extensive-stage small cell lung cancer: A multicentre, randomised, double-blind, placebo-controlled Phase II trial. Int J Cancer. 2021 May 15;148(10):2557-2570. doi: 10.1002/ijc.33453. Epub 2021 Jan 12. PMID 33348420
- [Background] Hart LL, Ferrarotto R, Andric ZG, Beck JT, Subramanian J, Radosavljevic DZ, Zaric B, Hanna WT, Aljumaily R, Owonikoko TK, Verhoeven D, Xiao J, Morris SR, Antal JM, Hussein MA. Myelopreservation with Trilaciclib in Patients Receiving Topotecan for Small Cell Lung Cancer: Results from a Randomized, Double-Blind, Placebo-Controlled Phase II Study. Adv Ther. 2021 Jan;38(1):350-365. doi: 10.1007/s12325-020-01538-0. Epub 2020 Oct 29. PMID 33123968
- [Background] Weiss J, Goldschmidt J, Andric Z, Dragnev KH, Gwaltney C, Skaltsa K, Pritchett Y, Antal JM, Morris SR, Daniel D. Effects of Trilaciclib on Chemotherapy-Induced Myelosuppression and Patient-Reported Outcomes in Patients with Extensive-Stage Small Cell Lung Cancer: Pooled Results from Three Phase II Randomized, Double-Blind, Placebo-Controlled Studies. Clin Lung Cancer. 2021 Sep;22(5):449-460. doi: 10.1016/j.cllc.2021.03.010. Epub 2021 Mar 26. PMID 33895103
- [Background] Lai AY, Sorrentino JA, Dragnev KH, Weiss JM, Owonikoko TK, Rytlewski JA, Hood J, Yang Z, Malik RK, Strum JC, Roberts PJ. CDK4/6 inhibition enhances antitumor efficacy of chemotherapy and immune checkpoint inhibitor combinations in preclinical models and enhances T-cell activation in patients with SCLC receiving chemotherapy. J Immunother Cancer. 2020 Oct;8(2):e000847. doi: 10.1136/jitc-2020-000847. PMID 33004541